CLINICAL TRIAL: NCT00711854
Title: Randomized Clinical Trial to Compare a Regimen of Trimethoprim-sulfamethoxazole (TMP-SMX) Plus Rifampicin With a Regimen of Linezolid in the Treatment of Infections Caused by Methicillin-resistant Staphylococcus Aureus (MRSA)
Brief Title: Randomized Clinical Trial to Compare a Regimen of Trimethoprim-sulfamethoxazole Plus Rifampicin With a Regimen of Linezolid in the Treatment of Methicillin-Resistant Staphylococcus Aureus (MRSA) Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Stephen Harbarth, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-059
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: MRSA Infection
Keywords: Staphylococcal infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Linezolid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): trimethoprim-sulfamethoxazole (TMP-SMX) plus rifampicin
  Interventions: Drug: trimethoprim-sulfamethoxazole (TMP-SMX); Drug: Rifampicin
- 2 (Active Comparator): Linezolid
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole (TMP-SMX) — TMP-SMX (160 mg TMP/ 800 mg SMX IV or PO 3x daily)
  Arms: 1
Drug: Linezolid — Linezolid (600 mg IV or PO twice daily)
  Arms: 2
Drug: Rifampicin — Rifampicin (600 mg IV or PO once daily)
  Arms: 1

SUMMARY:
MRSA infections often require systemic antibiotic therapy and represent an important healthcare burden. Currently available treatment options are either only available in parenteral form (vancomycin) or expensive (linezolid). Thus, there is an urgent, unmet need to better investigate in-expensive but highly active alternatives to currently recommended standard treatment options. The purpose of the proposed study is to test the hypothesis that a combination of TMP-SMX and rifampicin is not inferior to linezolid for treatment of MRSA infections.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients with clinical signs and symptoms of MRSA-related infection
3. Culture of MRSA (predominant microorganism in culture) susceptible to all of the following:

   * TMP-SMX
   * rifampicin
   * linezolid
4. Patient must give written informed consent to participate in the study.

Exclusion Criteria:

1. Women who are pregnant or nursing
2. Women who refuse to substitute oral contraception during treatment
3. Known or suspected hypersensitivity to linezolid, TMP-SMX or rifampicin
4. Clinical or laboratory evidence of significant impairment of hepatic function, as demonstrated by any of the following criteria:

   * Bilirubin > 3 x upper limit of normal range
   * AST or ALT > 5 x upper limit of normal range
   * Acute hepatitis or proven liver cirrhosis by liver histology
5. Treatment with other antimicrobials with activity against MRSA for > 72 hours prior to study inclusion
6. Patients with a high probability of death within the week following study entry
7. Patients who, in the opinion of the investigator, cannot be relied upon for post-therapy follow-up
8. Patients requiring alternative antibiotic therapy with anti-MRSA activity. However, if another antibiotic treatment without antistaphylococcal activity is necessary, the patient is acceptable for randomization. In that sense, the use of aztreonam (against Gram negative microorganisms) or metronidazole (against anaerobes) is allowed
9. Hemodialyzed patients
10. History of pheochromocytoma, carcinoid syndrome, untreated hyperthyroidism, uncontrolled hypertension, or patients receiving serotonin uptake inhibitors
11. Severe thrombocytopenia (< 50.000 platelets)
12. Left-sided endocarditis with a poor prognosis (patients aged over 50; cerebral embolism)
13. Chronic osteomyelitis without surgical debridement; superinfected indwelling foreign body, deliberately kept in place
14. Patients with severe sepsis or septic shock due to MRSA bacteremia
15. Patients who receive any of the following drugs, which cannot be substituted or temporarily withdrawn: adrenergic and serotonergic agents, tramadol, pethidine, duloxetine, venlafaxine, milnacipran, sibutramine, chlorpheniramine, brompheniramine, cyproheptadine, citalopram, and paroxetine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Bacteriological and clinical cure | 6 weeks

SECONDARY OUTCOMES:
Treatment costs | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Harbarth, MD, MS, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Harbarth S, von Dach E, Pagani L, Macedo-Vinas M, Huttner B, Olearo F, Emonet S, Uckay I. Randomized non-inferiority trial to compare trimethoprim/sulfamethoxazole plus rifampicin versus linezolid for the treatment of MRSA infection. J Antimicrob Chemother. 2015 Jan;70(1):264-72. doi: 10.1093/jac/dku352. Epub 2014 Sep 10. PMID 25209610
- See also: MRSA research center, Geneva University Hospitals and Medical School — http://medweb1.unige.ch/recherche/groupes/b_donnees/sujet_330_1.html